CLINICAL TRIAL: NCT02083042
Title: Clinical Validation of Lophius Biosciences Kit T-Track® CMV to Assess the Functionality of CMV-specific Cell-mediated Immunity (CMI) and Its Suitability to Determine a Protective Cut-off Value for CMV Reactivations/Disease in Kidney Transplant Recipients
Brief Title: Clinical Validation of Lophius Biosciences Kit T-Track® CMV in Kidney Transplant Recipients
Acronym: CMValue
Status: Completed | Type: Observational
Sponsor: Lophius Biosciences GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: LB-A2(Urea-CMV)
Record Dates: First submitted 2014-02-23; First posted 2014-03-11 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Cytomegalovirus; Kidney Transplantation; CMV Specific Immune Response
Keywords: CMV; T-Track CMV; kidney transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study aims to validate whether Lophius Biosciences Kit T-Track® CMV is suitable to assess the functionality of CMV-specific cell-mediated immunity (CMI) and to determine a protective cut-off value for CMV reactivations/disease in kidney transplant recipients.

Lophius kit T-Track® CMV represents a highly standardized and sensitive diagnostic tool to assess the functionality of a network of clinically relevant CMV-reactive effector cells. It is based on the stimulation of peripheral blood mononuclear cells (PBMC) with urea-formulated immunodominant CMV proteins, pp65 and IE-1, and the subsequent quantification of CMV-specific CMI (spot forming colonies) using a highly sensitive IFN-γ ELISpot.

DETAILED DESCRIPTION:
Severe clinical complications including acute rejection and opportunistic infections in solid organ transplantation (SOT) are mainly caused by inadequate impairment of cell-mediated immunity (CMI) by immunosuppressive therapy. In particular CMV is responsible for increased morbidity and mortality revealing the need for either prophylactic or preemptive antiviral treatment. Recipients with negative CMV serology (R-) receiving a graft from a seropositive donor (D+) are at highest risk of developing CMV-associated complications. Therefore, these patients usually receive antiviral prophylaxis whereas patients at intermediate risk (D+/R+ or D-/R+) are treated either prophylactically or preemptively. Although prophylaxis is efficient, it is also accompanied by harmful side effects and high costs. Thus, there is a need for a personalized antiviral as well as immunosuppressive therapy to optimally treat the patient and to improve long-term patient and graft survival. The detection of a protective threshold of functional CMV-reactive cells may help to predict the onset of viral complications, thereby minimizing harmful side effects. Currently available tools to measure CMV-specific cellular immunity reveal striking limitations including a lack of standardization necessitating a commercially available standardized test system. The Lophius kit T-Track® CMV represents a highly standardized and sensitive diagnostic tool to assess the functionality of a network of clinically relevant CMV-reactive effector cells. It is based on the stimulation of peripheral blood mononuclear cells (PBMC) with urea-formulated immunodominant CMV proteins, pp65 and IE-1, and the subsequent quantification of CMV-specific CMI (spot forming colonies) using a highly sensitive IFN-γ ELISpot. This study aims to assess the suitability of the Lophius Biosciences kit T-Track® CMV to determine the CMV-specific CMI in renal transplant recipients scheduled for a preemptive antiviral treatment strategy. Furthermore, it will be investigated if the results obtained with T-Track® CMV are suitable to define a cut-off value of CMV-specific CMI mediating protection from CMV reactivations and related complications. Moreover, possible associations between CMV-specific CMI measured with T-Track® CMV and clinical complications including acute rejection episodes and opportunistic infections will be analyzed as well as the influence of the immunosuppressive treatment and the patient's HLA type on viral immunity.

ELIGIBILITY:
Inclusion Criteria:

* Patient receiving a kidney graft
* Recipient being CMV-seropositive prior transplantation and receiving a graft from either a CMV-seropositive or from a seronegative donor (intermediate risk groups, D+/R+; D-/R+,)
* Patient scheduled to follow the preemptive antiviral strategy with oral valganciclovir or intravenous ganciclovir after transplantation
* Patient receiving the standard triple immunosuppressive regimen (CNI, MMF/MPA or mTOR inhibitors, steroids), with or without induction therapy (except ATG) as start therapy after transplantation
* Male or female patient at least 18 years of age
* Written informed consent

Exclusion Criteria:

* Patient is scheduled for the optional visit 1, but requires ongoing treatment with a systemic immunosuppressive drug already prior to kidney transplantation (except induction therapy other than ATG)
* Patient receiving ATG as induction therapy
* Patient is known to be positive for HIV or suffering from chronic hepatitis infections
* Patient has significant uncontrolled concomitant infections or other unstable medical conditions before transplantation that could interfere with the study objectives
* Patient is unable to comply with the visit schedule in the protocol
* Patient has any form of substance abuse, psychiatric disorder or condition that, in the opinion of the investigator may invalidate communication with the investigator

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Kidney transplant recipients of intermediate risk groups for CMV serostatus (D+/R+; D-/R+), and scheduled for the preemptive antiviral strategy
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2013-08; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Determination of changes in pp65 and/or IE-1 specific CMI applying T-Track® CMV | before Tx, week 3,6,9,12,15,18 and 21 after Tx and unscheduled visits in case of suspicion of CMV related complications; individual observation period 6 months

SECONDARY OUTCOMES:
Changes in CMV viral load measured by CMV-PCR or pp65 antigenemia test | week 3,6,9,12,15,18,21 after Tx and in case of CMV complications

OTHER OUTCOMES:
opportunistic infections, graft damage/rejection/loss, | 6 months after Tx

CONTACTS AND LOCATIONS:
Locations (1):
- Lophius Biosciences GmbH, Regensburg, Germany

REFERENCES:
- [Derived] Banas B, Steubl D, Renders L, Chittka D, Banas MC, Wekerle T, Koch M, Witzke O, Muhlfeld A, Sommerer C, Habicht A, Hugo C, Hunig T, Lindemann M, Schmidt T, Rascle A, Barabas S, Deml L, Wagner R, Kramer BK, Kruger B. Clinical validation of a novel enzyme-linked immunosorbent spot assay-based in vitro diagnostic assay to monitor cytomegalovirus-specific cell-mediated immunity in kidney transplant recipients: a multicenter, longitudinal, prospective, observational study. Transpl Int. 2018 Apr;31(4):436-450. doi: 10.1111/tri.13110. Epub 2018 Jan 16. PMID 29284181